CLINICAL TRIAL: NCT07369791
Title: A Phase II Study of Nivolumab Plus Relatlimab 360 mg/360 mg and Gemcitabine/Cisplatin as First-Line Treatment in Patients With Advanced Biliary Tract Cancer.(NOBLE）
Brief Title: Nivolumab Plus Relatlimab and Gemcitabine/Cisplatin as First-Line Treatment in Advanced Biliary Tract Cancer.
Acronym: NOBLE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); Tri-Service General Hospital (Other); National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1226
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer(BTC)
Keywords: Advanced Biliary Tract Cancer; randomization; chemoimmunotherapy
MeSH Terms: interventions — Nivolumab; Gemcitabine; Cisplatin; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab plus relatlimab 360 mg/360 mg in combination with GC (Experimental): Specified dose on specified days
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Nivolumab/Relatlimab
- Nivolumab in combination with GC (Active Comparator): Specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Arms: Nivolumab in combination with GC
Drug: Gemcitabine — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days
Drug: Nivolumab/Relatlimab — Specified dose on specified days
  Arms: Nivolumab plus relatlimab 360 mg/360 mg in combination with GC

SUMMARY:
A Randomized Phase II Study. To assess the difference in objective response rate (ORR) between adult patients with advanced biliary tract cancer assigned to nivolumab plus relatlimab 360 mg/360 mg in combination with GC or nivolumab plus GC as first-line treatment.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the difference in objective response rate (ORR) between adult patients with advanced biliary tract cancer assigned to nivolumab plus relatlimab 360 mg/360 mg in combination with GC or nivolumab plus GC as first-line treatment.

The primary endpoint will be evaluating ORR of nivolumab plus relatlimab 360 mg/360 mg in combination with gemcitabine and cisplatin in patients with advanced BTC.

A total of 76 evaluable subjects will be required for the study, where an evaluable subject is defined as a participant who has at least one post-treatment imaging assessment that is considered evaluable. To account for potential drop-outs or subjects without evaluable post-treatment imaging, the planned enrollment target is approximately 84 subjects, assuming an estimated 10% drop-out rate. After a participant's initial eligibility is established and informed consent has been obtained, the participant will be randomized in a 1:1 ratio to either the nivolumab + relatlimab + GC arm or the nivolumab + GC arm.

Randomization will be stratified by PD-L1 expression (combined positive score [CPS] ≥1 vs <1) and will be centrally assigned using a randomization table. Enrollment will not be restricted by evaluability at the time of registration; however, the number of evaluable subjects will be monitored throughout the trial. If the number of non-evaluable subjects exceeds the anticipated rate, additional participants may be enrolled to ensure that the target of 76 evaluable subjects is achieved.

Eligible patients will receive nivolumab 360 mg or nivolumab 360 mg plus relatlimab 360 mg on Day 1, along with gemcitabine 1000 mg/m² and cisplatin 25 mg/m² on Days 1 and 8 of each 3-week cycle.

Nivolumab and relatlimab will be administered for a maximum of 2 years. Cisplatin will be given for a maximum of 8 cycles. Gemcitabine will be given continuously until disease progression, intolerable toxicity, or patient withdrawal of consent at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed biliary tract carcinoma (including intrahepatic bile duct, extrahepatic bile duct, ampulla of Vater cancer, and gallbladder);
2. metastatic or unresectable disease;
3. no history of chemotherapy or radiotherapy or immunotherapy for biliary tract cancer, except for patients who experienced recurrence at least six months after completing adjuvant therapy;
4. presence of at least one measurable tumor lesion which is defined as lesions that can be accurately measured in at least 1 dimension with longest diameter (LD) ≥20 mm using conventional techniques or ≥10 mm with spiral CT and MRI; measurable lymph nodes must be ≥15 mm in the short axis;
5. must have PD-L1 testing with results performed by a local laboratory during the screening period
6. adequate hematopoietic function which is defined as below:

   1. hemoglobin level ≥ 9 g/dL;
   2. absolute neutrophil count (ANC) ≥ 1,500/mm3;
   3. platelet count ≥ 100,000/mm3;
7. adequate hepatic function which is defined as below:

   1. total bilirubin ≤ 2 times upper limit of normal (ULN);
   2. Alanine aminotransferase (ALT) ≤ 3 x ULN; if liver metastasis, ALT ≤ 5 x ULN
8. adequate renal function: creatinine clearance rate (CCr) ≥ 50 mL/min, calculated by Cockroft-Gault formula;< Cockroft-Gault formula > Male: ((140 - age) × weight [kg])/(72 × serum creatinine[mg/dL]) Female: 0.85 x estimate for male
9. age of 18 years or above
10. ECOG performance status 0-1;
11. life expectancy of at least 12 weeks;
12. ability to understand and willingness to sign a written informed consent document.
13. Subjects with chronic hepatitis B virus infection (HBV surface antigen (HBsAg) positive) must start antiviral therapy with nucleoside analogs (e.g., entecavir or tenofovir, according to current practice guidelines) before start of study drug treatment.

Exclusion Criteria:

1. other malignancy within the past 2 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ;
2. history or known presence of brain metastasis;
3. presence of grade 2 or above ascites or pleural effusion;
4. presence of grade 2 or above diarrhea;
5. presence of mental disease or psychotic manifestation;
6. active or uncontrolled infection;
7. Significant medical conditions that are contraindicated to study medication or render the patient at high risk from treatment complications, such as: Biliary tract-related infection or sepsis. Uncontrolled biliary obstruction. Ongoing grade ≥2 infection at any site despite appropriate therapy.;
8. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

   * Myocardial infarction (MI) or stroke/transient ischemic attack within the 6 months prior to consent
   * Uncontrolled angina within the 3 months prior to consent
   * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes or poorly controlled atrial fibrillation)
   * QTc prolongation > 480 msec
   * History of other clinically significant cardiovascular disease (ie, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc.)
   * Cardiovascular disease-related requirement for daily supplemental oxygen
   * History of 2 or more MIs OR 2 or more coronary revascularization procedures
   * Participants with history of myocarditis, regardless of etiology
   * Troponin T (TnT) or I (TnI) > 2 institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 × ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac evaluation and be considered for treatment, based on a favorable benefit-risk assessment by the Investigator.
9. Pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study and 5 months after treatment completion. Individuals of childbearing potential and male participants with a partner with childbearing potential should be counselled on the importance of pregnancy prevention and the potential of fetal toxicity occurring due to transmission of study intervention via seminal fluid to a developing fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1. Disease control is defined as having confirmed complete or partial response or stable disease for at least 12 weeks.
Duration of response (DOR) | Up to approximately 2 years
Progression-free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to 5 years
Safety profiles | Up to approximately 2 years
  Any toxicity other than hematology and biochemistry assessment shall be recorded and graded according to NCI-CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Huang Chen, MD, PhD, Study Director — Taipei Veterans General Hospital, Taiwan; Hui-Jen Tsai, MD, PhD, Principal Investigator — National Health Research Institutes, Taiwan; Chia-Jui Yen, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital; Shiue-Wei Lai, MD, PhD, Principal Investigator — Tri-Service General Hospital; Chiun Hsu, MD, PhD, Principal Investigator — National Taiwan University Hospital; Li-yuan Bai, MD, PhD, Principal Investigator — China Medical University Hospital; Yi-Chang Liu, MD, PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital; Nai-Wen Su, MD, Principal Investigator — Mackay Memorial Hospital; Hsin-Chen Lin, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (8):
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided